CLINICAL TRIAL: NCT01939366
Title: Efficacy, Safety and Tolerability of Multiple Doses of Oral Cebranopadol in Subjects With Moderate to Severe Chronic Pain Due to Diabetic Peripheral Neuropathy.
Brief Title: Cebranopadol Efficacy and Safety in Diabetic Patients Suffering From Chronic Pain Caused by Damage to the Nerves
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tris Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KF6005/08; 2013-000473-68 (EudraCT Number); U1111-1151-4331 (Other: WHO UTN)
Record Dates: First submitted 2013-09-06; First posted 2013-09-11 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain; Diabetic Neuropathies; Diabetes Mellitus
Keywords: Painful Diabetic Peripheral Neuropathy
MeSH Terms: conditions — Chronic Pain; Diabetic Neuropathies; Diabetes Mellitus | interventions — 6'-fluoro-4',9'-dihydro-N,N-dimethyl-4-phenylspiro(cyclohexane-1,1'(3'H)-pyrano(3,4-b)indol)-4-amine; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Cebranopadol 300 µg (Experimental)
  Interventions: Drug: Cebranopadol 300 µg
- Cebranopadol 600 µg (Experimental)
  Interventions: Drug: Cebranopadol 600 µg
- Pregabalin (Active Comparator)
  Interventions: Drug: Pregabalin
- Matching Placebo (Placebo Comparator)
  Interventions: Drug: Matching Placebo
- Cebranopadol 100 µg (Experimental)
  Interventions: Drug: Cebranopadol 100 µg

INTERVENTIONS:
Drug: Cebranopadol 100 µg — Participants randomized to 100 μg cebranopadol will start with 100 μg per day and will remain on 100 µg per day.
  Arms: Cebranopadol 100 µg
Drug: Cebranopadol 300 µg — Participants randomized to 300 μg cebranopadol will start with 100 μg per day and increase to 300 µg per day on day 4 and will remain on 300 µg per day.
  Arms: Cebranopadol 300 µg
Drug: Cebranopadol 600 µg — Participants randomized to 600 μg cebranopadol will start with 200 μg per day and increase to 400 µg per day on day 4 and to 600 µg on day 7, thereafter they will remain on 600 µg per day.
  Arms: Cebranopadol 600 µg
Drug: Pregabalin — Stepwise titration from 75 mg twice a day to 300 mg twice a day over 2 weeks.
  Other Names: Lyrica®
  Arms: Pregabalin
Drug: Matching Placebo — Placebo will be matched to pregabalin and cebranopadol.
  Arms: Matching Placebo

SUMMARY:
The purpose of this trial is to evaluate if cebranopadol is safe and can decrease pain in patients when compared to placebo (a tablet that does not contain active product) and when compared to a marketed product containing pregabalin (Lyrica®). Furthermore, this trial will be undertaken to find out if the patient's general health and well-being improves under trial treatment.

The concentrations of cebranopadol in the blood will be investigated to get a better understanding of how it is absorbed from the gut, distributed and broken down in the body, and eliminated from the body.

ELIGIBILITY:
Inclusion Criteria:

* written signed informed consent
* type 1 or type 2 diabetes mellitus
* clinical diagnosis of painful Diabetic Polyneuropathic Neuropathy (DPN) with symptoms and signs for at least 3 months
* must require medication (e.g., non-opioids or opioids up to an equivalent dose of 160 mg oral morphine/day) for the treatment of pain due to DPN for at least 1 month prior to Visit 1 and must be dissatisfied with the current treatment (in terms of efficacy and/or tolerability). Medication for the treatment of pain due to DPN should be required on at least 4 of 7 consecutive days.
* blood glucose to be controlled by a diet, oral anti-hyperglycemic medication, and/or insulin for at least 3 months prior. Glycosylated hemoglobin (HbA1C) should not be greater than 11%
* baseline pain intensity score greater or equal to 5 on the 11-point Numerical Rating Scale (NRS) without intake of any analgesic at allocation. For each of the last 3 days prior to allocation of treatment, a 24 hour NRS score greater or equal to 4 is required
* women of childbearing potential must have a negative urine pregnancy test at enrollment
* using medically acceptable and highly effective methods of birth control (and willing to use them during the trial).

Exclusion Criteria:

* presence of other pain that could confound the painful Diabetic Polyneuropathy (DPN) assessments, e.g. pain due to nerve entrapment (tarsal tunnel syndrome, osteoarthritis of the knee etc), peripheral vascular disease, radiculopathy, plantar fasciitis, tendonitis, mononeuritis multiplex, postherpetic neuralgia, complex regional pain syndrome, or fibromyalgia.
* neuropathy due to etiologies other than diabetes, e.g. autoimmune disorders, inflammatory neuropathies (e.g. chronic inflammatory demyelinating polyneuropathy), thyroid disease or endocrine disorders (other than diabetes), heavy metal or toxic neuropathy, nutritional deficiency, metabolic disorders, vasculitis, infections, injury, or paraneoplastic syndromes.
* severe or extensive diabetic ulcers or amputations due to diabetes
* Charcot's joints due to diabetes.
* any clinically significant disease or laboratory findings, e.g., significant unstable cardiac, vascular, pulmonary, gastrointestinal, endocrine, metabolic, neurological, or psychiatric disorders.
* inability to comply with the protocol and with the intake of trial medication that, in the investigator's opinion, might indicate that the participant is unsuitable for the trial.
* conditions that require treatment with medication that is not allowed to be taken during the trial
* previous or current alcohol or drug abuse or opioid dependency.
* severe functional hepatic impairment corresponding to Child-Pugh classification C.
* history of acute hepatitis
* impaired renal function, a creatinine clearance less than 60 mL/min at the enrollment (Cockcroft-Gault calculated).
* history of any major gastrointestinal procedures (e.g., gastric bypass) or gastrointestinal conditions (e.g. acute diarrhea, blind loop syndrome, gastric dumping syndrome, Whipple's disease) that might affect the absorption or metabolism of cebranopadol or pregabalin.
* risk factors for or history of torsade de pointes and/or marked prolongation of the QT interval (e.g. heart failure, hypokalemia, or bradycardia).
* history of seizure disorder and/or epilepsy or any condition associated with a significant risk for seizure disorder or epilepsy at the discretion of the investigator.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2013-09-27 (Actual); Primary Completion 2015-01 (Actual); Study Completion 2015-01-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Director Clinical Trials, Study Director — Grünenthal GmbH
Locations (82):
- United States (15):
  - US002, Mesa, Arizona
  - US001, Garden Grove, California
  - US019, Laguna Hills, California
  - US014, National City, California
  - US007, Orange, California
  - US011, Hialeah, Florida
  - US012, Miami, Florida
  - US009, Orlando, Florida
  - US004, Blackfoot, Idaho
  - US006, Elgin, Illinois
  - US016, West Long Branch, New Jersey
  - US008, Brooklyn, New York
  - US005, Brooklyn, New York
  - US021, New York, New York
  - US003, West Jordan, Utah
- Austria (7):
  - AT007, Graz
  - AT005, Salzburg
  - AT004, Senftenberg
  - AT002, Vienna
  - AT003, Vienna
  - AT001, Vienna
  - AT006, Vienna
- Denmark (4):
  - DK005, Aalborg
  - DK003, Aarhus
  - DK002, Copenhagen
  - DK001, Odense
- France (7):
  - FR008, Corbeil-Essonnes
  - FR001, Lille
  - FR007, Limoges
  - FR005, Montauban
  - FR002, Nantes
  - FR004, Orléans
  - FR006, Paris
- Germany (31):
  - DE018, Aschaffenburg
  - DE003, Bad Oeynhausen
  - DE005, Berlin
  - DE023, Berlin
  - DE031, Berlin
  - DE004, Berlin
  - DE025, Berlin
  - DE013, Bochum
  - DE033, Dresden
  - DE017, Düsseldorf
  - DE012, Düsseldorf
  - DE010, Essen
  - DE034, Essen
  - DE022, Essen
  - DE006, Frankfurt
  - DE007, Görlitz
  - DE021, Hamburg
  - DE020, Hanover
  - DE016, Karlsruhe
  - DE002, Kiel
  - DE030, Künzing
  - DE008, Leipzig
  - DE009, Leipzig
  - DE015, Magdeburg
  - DE032, Magdeburg
  - DE001, Mainz
  - DE028, Mayen
  - DE027, München
  - DE014, Münster
  - DE011, Neuss
  - DE024, Schwerin
- Italy (4):
  - IT005, Ancona
  - IT004, Milan
  - IT001, Rome
  - IT002, Turin
- Netherlands (8):
  - NL007, Amsterdam
  - NL004, Apeldoorn
  - NL005, Beek
  - NL001, Eindhoven
  - NL002, Rotterdam
  - NL006, Venlo
  - NL008, Zwijndrecht
  - NL003, Zwolle
- Spain (6):
  - ES001, Cuenca
  - ES011, Madrid
  - ES010, Madrid
  - ES009, Madrid
  - ES003, Toledo
  - ES006, Valencia

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The trial started on 27 Sep 2013 with the enrollment of the first participants and was completed on 28 Jan 2015 when the last participant completed the last follow-up examination according to the protocol.
Pre-assignment Details: Of the 699 participants enrolled 370 participants were not allocated (322 did not meet the eligibility criteria, 29 withdrew consent, 6 due to Adverse Events, 2 due to protocol deviations, 11 due to other reasons). 13 participants allocated to treatment were excluded from the PPS, FAS & SAF analyses populations due to GCP non-compliance at 2 sites.
Period: Overall Study
Arm/Group | Cebranopadol 100 µg | Cebranopadol 300 µg | Cebranopadol 600 µg | Pregabalin | Matching Placebo
Started | 66 | 64 | 65 | 68 | 66
Allocated Set Excl. Non-compliant Sites | 64 | 61 | 63 | 65 | 63
Safety Set | 64 | 61 | 62 | 65 | 62
Full Analysis Set | 64 | 60 | 61 | 65 | 62
Per Protocol Set | 58 | 55 | 50 | 51 | 49
Completed | 52 | 41 | 27 | 51 | 48
Not Completed | 14 | 23 | 38 | 17 | 18
Not completed — Adverse Event | 8 | 17 | 30 | 8 | 5
Not completed — Lack of Efficacy | 2 | 1 | 1 | 1 | 3
Not completed — Lost to Follow-up | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 2 | 2 | 3
Not completed — Inclusion criteria not met | 0 | 1 | 1 | 0 | 1
Not completed — Other | 0 | 0 | 2 | 2 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0
Not completed — Sponsor decision | 0 | 0 | 0 | 0 | 2
Not completed — GCP non-compliance at site | 2 | 3 | 2 | 3 | 3

BASELINE CHARACTERISTICS:
Population: Full Analysis Set
Groups:
- Total: Total of all reporting groups
Arm/Group | Cebranopadol 100 µg | Cebranopadol 300 µg | Cebranopadol 600 µg | Pregabalin | Matching Placebo | Total
Number analyzed (Participants) | 64 | 61 | 62 | 65 | 62 | 314
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.2 (8.6) | 61.6 (8.7) | 62.2 (8.1) | 61.7 (9.9) | 63.3 (10.3) | 62.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 23 | 22 | 16 | 13 | 94
  Male | 44 | 38 | 40 | 49 | 49 | 220
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 7 | 6 | 6 | 10 | 5 | 34
  Not Hispanic or Latino | 57 | 55 | 56 | 55 | 57 | 280
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 1 | 0 | 0 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 0 | 2 | 4 | 1 | 9
  White | 61 | 58 | 57 | 58 | 61 | 295
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 2 | 3 | 0 | 6
Region of Enrollment [Number; unit: participants]
  Austria | 5 | 6 | 5 | 6 | 5 | 27
  Netherlands | 3 | 3 | 4 | 2 | 4 | 16
  United States | 13 | 10 | 9 | 13 | 10 | 55
  Denmark | 2 | 2 | 2 | 1 | 2 | 9
  Italy | 2 | 2 | 2 | 2 | 1 | 9
  France | 7 | 7 | 8 | 8 | 8 | 38
  Germany | 31 | 30 | 30 | 32 | 31 | 154
  Spain | 1 | 1 | 2 | 1 | 1 | 6
Height [Mean (Standard Deviation); unit: meter] | 1.721 (0.098) | 1.736 (0.092) | 1.717 (0.104) | 1.736 (0.110) | 1.736 (0.076) | 1.729 (0.097)
Weight [Mean (Standard Deviation); unit: kilogram] | 95.77 (15.62) | 96.51 (18.12) | 93.72 (16.05) | 92.25 (17.28) | 99.00 (15.99) | 95.42 (16.69)
BMI [Mean (Standard Deviation); unit: kilogram per square meter] | 32.30 (4.41) | 31.87 (4.39) | 31.70 (4.29) | 30.66 (5.26) | 32.80 (4.53) | 31.86 (4.62)
Pain Assessment - Average 24-hour pain [Mean (Standard Deviation); unit: units on a scale] — Participants recorded their current pain twice daily (morning and evening), and, with a recall period of 24 hours, their worst and 24-hour pain once daily in the evening. Pain was assessed using an 11-point numerical rating scale (NRS). Participants had to select a number corresponding to their pain, with anchors at 0 for "no pain" and 10 for "pain as bad as you can imagine". The average baseline pain was calculated as the average over the three 24-hour pain assessments of the last 3 days prior to the Baseline Visit.
  units on a scale | 6.92 (1.34) | 6.80 (1.37) | 6.80 (1.25) | 6.78 (1.22) | 6.84 (1.15) | 6.83 (1.26)
Pain Assessment - Worst 24-hour pain [Mean (Standard Deviation); unit: units on a scale] — Participants recorded their current pain twice daily (morning and evening), and, with a recall period of 24 hours, their worst and 24-hour pain once daily in the evening. Pain was assessed using an 11-point numerical rating scale (NRS). Participants had to select a number corresponding to their pain, with anchors at 0 for "no pain" and 10 for "pain as bad as you can imagine". The worst 24-hour pain was calculated as the average over the three 24-hour pain assessments of the last 3 days prior to the Baseline Visit.
  units on a scale | 7.41 (1.36) | 7.32 (1.28) | 7.38 (1.21) | 7.32 (1.16) | 7.33 (1.14) | 7.35 (1.23)
Pain Assessment - Current Morning Pain [Mean (Standard Deviation); unit: units on a scale] — Participants recorded their current pain twice daily (morning and evening), and, with a recall period of 24 hours, their worst and 24-hour pain once daily in the evening. Pain was assessed using an 11-point numerical rating scale (NRS). Participants had to select a number corresponding to their pain, with anchors at 0 for "no pain" and 10 for "pain as bad as you can imagine". The current morning pain at baseline was calculated as the average over the three pain assessments of the last 3 days prior to the Baseline Visit.
  units on a scale | 6.60 (1.58) | 6.58 (1.53) | 6.44 (1.46) | 6.61 (1.44) | 6.58 (1.48) | 6.56 (1.49)
Pain Assessment - Current Evening Pain [Mean (Standard Deviation); unit: units on a scale] — Participants recorded their current pain twice daily (morning and evening), and, with a recall period of 24 hours, their worst and 24-hour pain once daily in the evening. Pain was assessed using an 11-point numerical rating scale (NRS). Participants had to select a number corresponding to their pain, with anchors at 0 for "no pain" and 10 for "pain as bad as you can imagine". The current evening pain at baseline was calculated as the average over the three pain assessments of the last 3 days prior to the Baseline Visit.
  units on a scale | 6.98 (1.50) | 6.87 (1.46) | 6.68 (1.33) | 6.75 (1.36) | 6.55 (1.34) | 6.80 (1.40)

OUTCOME MEASURES:

1. Primary Outcome: Change in Average Pain Intensity.
Description: Participants will be asked to record their pain intensity in the evening. Participants are asked to rate how much pain they had on average in the past 24 hours. The participant scores their pain intensity on an 11-point Numerical Rating Scale (NRS) where a score of 0 indicated "no pain" and a score of 10 indicated "pain as bad as you can imagine". Baseline average pain scores are calculated from the averages of all scores recorded during the 3 days prior to randomization. The average pain at week 6 will be the average pain scores calculated from all pain scores measured during week 6.
Time Frame: Baseline; to End of Week 6 of the Maintenance Phase
Population: Full Analysis Set (FAS). Mixed-effects model for repeated measures (MMRM).
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Cebranopadol 100 µg | Cebranopadol 300 µg | Cebranopadol 600 µg | Pregabalin | Matching Placebo
Number analyzed (Participants) | 64 | 60 | 58 | 64 | 61
units on a scale | -2.24 [-2.78 to -1.70] | -2.28 [-2.86 to -1.71] | -2.56 [-3.20 to -1.91] | -2.79 [-3.33 to -2.26] | -1.55 [-2.10 to -1.00]
Statistical Analysis 1: Comparison: Cebranopadol 100 µg vs Matching Placebo; The mixed model repeated measurement (MMRM) model included fixed effects of pooled sites, treatment, week, treatment-by-week interaction, baseline pain, and a subject-specific random effect. The model was based on the weekly average 24-hour pain intensity of the 2 weeks in the Titration Phase and 6 weeks in the Maintenance Phase. An unstructured covariance matrix was used to model the covariance structure, denominator degrees of freedom were estimated using the Kenward-Roger approximation; Test type: Superiority or Other; p = 0.0621, Mixed Models Analysis — Due to the exploratory character of this trial, no multiple testing adjustment for control of the false positive rate was applied; The analysis consisted of the contrasts (mixed model Wald tests) of individual cebranopadol doses versus placebo during Week 6 of Maintenance Phase; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.43 to 0.04], Standard Error of Mean 0.37
Statistical Analysis 2: Comparison: Cebranopadol 300 µg vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0564, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.74, 95% CI 2-sided [-1.50 to 0.02], Standard Error of Mean 0.39
Statistical Analysis 3: Comparison: Cebranopadol 600 µg vs Matching Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.0153, Mixed Models Analysis — [p-value comment as in outcome 1, analysis 1]; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-1.83 to -0.20], Standard Error of Mean 0.41

ADVERSE EVENTS:
Time Frame: Safety Analysis Set Baseline Visit (Day 1) to End of Maintenance Phase (Day 57).
Arm/Group | Cebranopadol 100 µg | Cebranopadol 300 µg | Cebranopadol 600 µg | Pregabalin | Matching Placebo
All-Cause Mortality (participants affected / at risk) | 0/64 | 0/61 | 0/62 | 0/65 | 0/62
Serious Adverse Events (participants affected / at risk) | 1/64 | 2/61 | 4/62 | 1/65 | 2/62
Other Adverse Events (participants affected / at risk) | 47/64 | 50/61 | 53/62 | 49/65 | 43/62
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cebranopadol 100 µg (N=64) | Cebranopadol 300 µg (N=61) | Cebranopadol 600 µg (N=62) | Pregabalin (N=65) | Matching Placebo (N=62)
Abdominal Pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 1
Diverticulum Intestinal Haemorrhagic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0 | 0
Peripheral Swelling (General disorders) | 0 | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Diabetes Mellitus (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0
Hypoglycaemic Coma (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Renal Failure Acute (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0
Haematoma (Vascular disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cebranopadol 100 µg (N=64) | Cebranopadol 300 µg (N=61) | Cebranopadol 600 µg (N=62) | Pregabalin (N=65) | Matching Placebo (N=62)
Abdominal pain upper (Gastrointestinal disorders) | 0 | 6 | 0 | 0 | 2
Constipation (Gastrointestinal disorders) | 3 | 6 | 7 | 6 | 2
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 3 | 2 | 5
Dry mouth (Gastrointestinal disorders) | 1 | 1 | 8 | 1 | 1
Nausea (Gastrointestinal disorders) | 6 | 22 | 16 | 6 | 6
Vomiting (Gastrointestinal disorders) | 2 | 10 | 17 | 1 | 2
Fatigue (General disorders) | 8 | 11 | 10 | 5 | 2
Oedema peripheral (General disorders) | 3 | 3 | 1 | 6 | 1
Bacteriuria (Infections and infestations) | 5 | 3 | 3 | 6 | 6
Nasopharyngitis (Infections and infestations) | 3 | 1 | 1 | 5 | 6
Weight increased (Investigations) | 0 | 0 | 0 | 5 | 1
Dizziness (Nervous system disorders) | 8 | 10 | 21 | 12 | 6
Headache (Nervous system disorders) | 3 | 6 | 3 | 4 | 2
Somnolence (Nervous system disorders) | 3 | 8 | 8 | 3 | 1
Tremor (Nervous system disorders) | 1 | 1 | 1 | 4 | 0
Depressed mood (Psychiatric disorders) | 1 | 1 | 2 | 0 | 4
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 3 | 8 | 6 | 1 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to review any proposed presentation of the results of this trial before they are submitted for publication or public disclosure. Neither party has the right to prohibit publication or public disclosure unless it can be shown to affect possible patent rights.